CLINICAL TRIAL: NCT06303648
Title: A Single, Ascending Dose Evaluation of the Safety, Pharmacokinetics of Methylone in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Transcend Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TSND201-PK-101
Record Dates: First submitted 2024-02-20; First posted 2024-03-12 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — methylone

STUDY DESIGN:
Intervention Model Description: Subjects will be enrolled into one of four cohorts. The study will begin enrolling Cohort 1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Cohort 1 (Experimental): 50 mg x 1 dose
  Interventions: Drug: Methylone
- Cohort 2 (Experimental): 100 mg x 1 dose
  Interventions: Drug: Methylone
- Cohort 3 (Experimental): 150 mg x 1 dose
  Interventions: Drug: Methylone
- Cohort 4 (Experimental): 200 mg x 1 dose
  Interventions: Drug: Methylone
- Cohort 5 (Experimental): 150 mg + 100 mg x 1
  Interventions: Drug: Methylone; Drug: Placebo

INTERVENTIONS:
Drug: Methylone — Oral dose of methylone
Drug: Placebo — Placebo to match methylone
  Arms: Cohort 5

SUMMARY:
This is an open-label, single, ascending dose study evaluating the PK and safety of methylone in healthy subjects.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy adult male or female aged 25 to 55 inclusive
* Normal resting ECG
* Normal hematologic and hepatic function
* Normal renal function

Key Exclusion Criteria:

* Vital sign abnormalities
* Positive urine drug screen at screening and / or Day -1
* Current mental illness such as depression, anxiety disorder, schizophrenia or other psychotic disorders

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-07-13 (Actual); Study Completion 2025-07-13 (Actual)

PRIMARY OUTCOMES:
Cmax: Maximum Observed Plasma Concentration for methylone | 48 hours following the dose
AUC: Area under the plasma concentration-time curve for methylone | 48 hours following the dose

SECONDARY OUTCOMES:
Incidence and frequency of adverse events | 10 days after the dose

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX Clinical Research, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No